CLINICAL TRIAL: NCT07371923
Title: Application of Zanubrutinib-based Combination Regimens in the Treatment of Newly-diagnosed Diffuse Large B-cell Lymphoma: A Phase II, Prospective, Single-center, Single-arm Clinical Study
Brief Title: Application of Zanubrutinib-based Combination Regimens in the Treatment of Newly-diagnosed Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, LIANG WANG, Director of department of hematology, Beijing Tongren Hospital, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRhos-DLBCL-01
Record Dates: First submitted 2025-11-18; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: diffuse large b cell lymphoma (DLBCL); BTK inhibitors; zanubrutinib; high-risk factors
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (for DLBCL patients witout central nervous system lesions) (Experimental): zanubrutinib combined with Pola-R-CHP regimen: zanubrutinib 160mg bid d1-d21/C1-C6; polatuzumab 1.8mg/kg d1/C1-C6; rituximab 375mg/㎡, iv, d1/C1-C6; cyclophosphamide 750mg/㎡, iv, d1/C1-C6; doxorubicin 50mg/㎡, iv, d1/C1-C6; predinisone 60mg/㎡ d1-5/C1-C6.
  Interventions: Drug: Zanubrutinib+Pola-R-CHP

INTERVENTIONS:
Drug: Zanubrutinib+Pola-R-CHP — zanubrutinib combined with Pola-R-CHP regimen: zanubrutinib 160mg bid d1-d21/C1-C6; polatuzumab 1.8mg/kg d1/C1-C6; rituximab 375mg/㎡, iv, d1/C1-C6; cyclophosphamide 750mg/㎡, iv, d1/C1-C6; doxorubicin 50mg/㎡, iv, d1/C1-C6; predinisone 60mg/㎡ d1-5/C1-C6.

SUMMARY:
Diffuse large B-cell lymphoma (DLBCL) is the most common type of non-Hodgkin's lymphoma. Currently, the first-line treatment regimen based on R-CHOP can only achieve clinical cure for 50% to 60% of patients. Previous studies have shown that patients with high-risk factors have a poor response to R-CHOP treatment and need further improvement. These high-risk factors include: IPI score ≥2 points, ABC subtype, double-expressing lymphoma, double-hit lymphoma, CD5-positive DLBCL, MCD subtype, N1 subtype, A53 subtype, extranodal lesions ≥2, special site involvement, such as central nervous system CNS, breast, testis, ovary, uterus, bone marrow, vitreoretinal, paraspinal, paranasal sinuses and intravascular, etc. Patients with DLBCL accompanied by high-risk factors also have a significantly increased risk of secondary CNS infiltration during recurrence. In previous RCHOP+X research strategies, only the combination of polatuzumab achieved significant 2-year PFS benefits in the overall population. None of the other studies achieved significant PFS benefits in the overall population. Therefore, the latest version of the CSCO guidelines recommends the Pola-R-CHP regimen as the first-line treatment for primary DLBCL. However, there is still considerable room for improvement in the survival of DLBCL patients with high-risk factors in clinical practice. Therefore, the strategy of the Pola-R-CHP-based combined with X regimen in high-risk DLBCL patients with specific risk factors can be explored subsequently.

The Phoenix study for young double expression of lymphoma patients, R - CHOP combined with BTK inhibitors can significantly improve the patient's survival, the subsequent omics data analysis indicates that MCD subtype, N1 subtypes and BN2 subtype can significantly benefit from BTK inhibitors. In addition, given that the proportion of MCD subtypes is high in most extranodal DLBCL patients and secondary CNS involvement is prone to occur, BTK inhibitors can effectively penetrate the blood-brain barrier (BBB) and have both preventive and therapeutic effects on CNS lesions. Therefore, exploring the application of BTK inhibitor zanubrutinib combined with R-CHOP or Pola-R-CHP regimens in high-risk DLBCL patients with specific risk factors (or zanubrutinib combined with rituximab and high-dose MTX in primary central nervous system DLBCL) has good application prospects. It is conducive to further improving the prognosis of such high-risk patients. Therefore, this study aimed to explore the efficacy and safety of the BTK inhibitor zanubrutinib combined with Pola-R-CHP regimen (or zanubrutinib combined with rituximab and high-dose MTX in primary central nervous system DLBCL, etc.) in patients of DLBCL with specific risk factors (IPI score two points or more, ABC subtypes, double expressor lymphoma, double hit lymphoma, CD5 positive DLBCL, MCD subtypes, N1 subtypes, A53 subtypes, extranodal lesions of 2 or more, special locations involved, such as the central nervous system (CNS, breast, testes).

DETAILED DESCRIPTION:
This study aimed to explore the efficacy and safety of the BTK inhibitor zanubrutinib combined with Pola-R-CHP regimen (or zanubrutinib combined with rituximab and high-dose MTX in primary central nervous system DLBCL, etc.) in patients of DLBCL with specific risk factors (IPI score two points or more, ABC subtypes, double expressor lymphoma, double hit lymphoma, CD5 positive DLBCL, MCD subtypes, N1 subtypes, A53 subtypes, extranodal lesions of 2 or more, special locations involved, such as the central nervous system (CNS, breast, testes).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diffuse large B-cell lymphoma (DLBCL);
* Have a "measurable lesions" ;
* Have at least one of the following risk factors, including: IPI score ≥2 points, ABC subtype, double-expressor lymphoma, double-hit lymphoma, CD5-positive DLBCL, MCD subtype, N1 subtype, A53 subtype, extranodal lesions ≥2, special site involvement, such as central nervous system CNS, breast, testis, ovary, uterus, bone marrow, vitreoretinal, paraspinal, paranasal sinuses and intravascular, etc.
* ECOG score 0-3;
* Expected survival time for 3 months or more;
* White blood cell count ≥3 x 10e9/L, the platelet count≥50 x 10e9/L; 1.5 mg/dL or less of serum creatinine, creatinine clearance≥50 ml/min; ALT, AST 3 x ULN or less, total bilirubin 2 x ULN or less.

Exclusion Criteria (the subject should not have any one of the following):

* currently suffering from other malignant tumor;
* ever received any treatments for lymphoma, except for short-term use of corticosteroids;
* Allergic to any kind of study drug;
* Active infection or uncontrol of HBV infection, HIV/AIDS or other serious infectious diseases;
* Pregnancy and lactation women of childbearing age and are reluctant to take contraception subjects;
* Researchers think that the subject does not fit to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Best complete remission rate (CRR) | From the start of the first cycle of treatment up to 24 weeks (when all six cycles of treatment was completed)
  Response assessment was done after every two cycles of treatment. Best CRR was defined as the CRR during all the six cycles of treatment.

SECONDARY OUTCOMES:
best overall response rate (ORR) | From the start of the first cycle of treatment up to 24 weeks (when all six cycles of treatment was completed).
  Response assessment was done after every two cycles of treatment. Best ORR was defined as the ORR during all the six cycles of treatment.
Two-year progression free survival (PFS) rate | From the start of the first cycle of treatment up to 24 months after initiation of treatment for the last enrolled patient.
  PFS was caculated from the date of start of treatment to date of disease progression, death of any cause, or last follow-up, whichever came first.
Two-year overall survival (OS) rate | From the start of the first cycle of treatment up to 24 months after initiation of treatment for the last enrolled patient.
  OS was caculated from the date of start of treatment to date of death of any cause, or last follow-up, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No